CLINICAL TRIAL: NCT02475291
Title: Clinical Usefulness of Fractional Flow Reserve Measurement for Significant Stenosis in Proximal Coronary Artery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2015-0025
Record Dates: First submitted 2015-06-08; First posted 2015-06-18 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease; Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Significant coronary lesions: Significant lesions with more than 70% diameter stenosis at proximal major coronary arteri(es).

SUMMARY:
Fractional flow reserve (FFR) is a pressure-wire-based index that is used during coronary angiography to assess the potential of a coronary stenosis to induce myocardial ischemia. Recent ESC guidelines referred to the usefulness of FFR extensively when noninvasive stress imaging is contraindicated, non-diagnostic, or unavailable. However, FFR requires additional manipulation with maximal and stable hyperemia by intravenous adenosine. More routine use of FFR for all angiographically significant stenoses would add considerable time, cost, and complexity to each PCI procedure and might also increase the risk of catheter-related complications such as coronary dissection and perforation. Although the guideline mentioned that FFR may not be useful in very high grade lesions (angiographically >90%) which always have an FFR <0.80, it have not been revealed yet proper criteria to predict FFR <0.80 obtained by angiographic parameters including degree of stenosis, lesion location and vessel size. It would be valuable to find more precise criteria available by conventional angiography for discrimination of functional stenosis in way to reduce the risk of additional procedure. For the purpose, the investigators will perform FFR in the lesions with significant stenosis (>70% diameter stenosis by visual estimation) and compare the angiographic parameters and FFR values in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Typical angina
* Stable or unstable angina pectoris
* At least one or more major epicardial coronary arteries with significant stenosis (>70% diameter stenosis by visual estimation on angiogram) confined to the proximal portion of left anterior descending artery, left circumflex artery, or right coronary artery
* Reference vessel diameter of target lesion ≥3.0 mm
* Normal LV ejection fraction (≥50%) without wall motion abnormality by echocardiography

Exclusion Criteria:

* Previous myocardial infarction
* Previous coronary bypass graft surgery
* Cardiogenic shock
* Multiple lesions in the vessel of interest
* Contraindication or hypersensitivity to adenosine or contrast media
* Reduced coronary blood flow (TIMI flow grade <3) in the vessel of interest
* Heavy calcified (definite calcified lesions on angiogram) or extremely tortuous lesions
* Pregnant women or women with potential childbearing
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant lesions with more than 70% diameter stenosis at proximal part of one or more major coronary arteries, regardless of revascularization strategy.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Agreement of diagnosis between FFR-documented ischemia and angiographically significant stenosis | 1day
  Coronary lesions with FFR <0.80 will be defined to be related with ischemia. Because all lesions in the study will be angiographically significant stenosis with DS >70%, agreement of diagnosis between FFR-defined ischemia and angiographically significant stenosis will be obtained by the ratio of lesions with FFR <0.80.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea